CLINICAL TRIAL: NCT02583295
Title: The Impact of Maternal Sound on Awareness for Pediatric Patients Undergoing Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sayed Kaoud Abd-Elshafy, Associate Professor (Anesthesiology and Critical Care)- College of Medicine, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB000087135
Record Dates: First submitted 2015-10-10; First posted 2015-10-22 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Intraoperative Awareness
Keywords: Awareness; Cardiac Surgery; Maternal; Pediatric; Sound; Music
MeSH Terms: conditions — Intraoperative Awareness

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Music group (Active Comparator): Music sound
  Interventions: Behavioral: Music sound
- Maternal sound group (Active Comparator): Maternal sound
  Interventions: Behavioral: Maternal sound

INTERVENTIONS:
Behavioral: Music sound — The recorded preferred songs or music (commercially available) listened by CD player connected to the patient ears before induction of anesthesia and continued during intra operative period
  Arms: Music group
Behavioral: Maternal sound — The recorded maternal voice (while they are singing the most popular songs their children like or telling a story to help their children to sleep) listened by CD player connected to the patient ears before induction of anesthesia and continued during intra operative period
  Arms: Maternal sound group

SUMMARY:
Awareness during anesthesia with intraoperative memory occurs when the patient is able to process information and produce specific responses to several stimuli. Anecdotal evidence suggests that children exposed to therapeutic suggestion consisting of gently encouraging, positive words spoken to them during emergence from anesthesia seem to arouse after surgery with less agitation, less pain and lower requirements for pain medications. Therapeutic suggestion has been associated with positive results in some adults during surgery, but it is unknown how therapeutic suggestion affects children. A newborn's recognition and preference for their mother's voice occurs early in life, very likely during fetal development. Additional evidence, revealed that at least as early as 4 months of age, infants process auditory stimuli from their mother's voice at a higher amplitude than they process auditory input from female strangers, suggesting that maternal voice stimuli undergo a unique form of cerebral processing that lends support for the existence of neurophysiologic mechanisms that reflect a child's preference for his/her mother's voice. This study aims to evaluate and compare the possibility of intra-operative awareness prevention by using either music listening or maternal sound listening in children undergoing cardiac surgery.

DETAILED DESCRIPTION:
children (4 to 8 years) undergoing repair of Atrial Septal Defect (ASD). Patients will be randomized into two groups (music group and maternal sound group); in music group patients listened to a recorded CD by music and songs preferred by the child, while in maternal sound group patients listened to a recorded CD where the mother singing the most popular songs their children like or telling a story to their children. In both groups bi spectral index (BIS) to detect depth of anesthesia. An interview will be conducted with the patients and their parent within the first postoperative week by a semi-structured in-depth questionnaire to evaluate occurrence of awareness.

ELIGIBILITY:
Inclusion Criteria:

* patients in the age range 4-8 years scheduled for elective cardiac surgery for Atrial Septal Defect (ASD) repair with Cardiopulmonary bypass

Exclusion Criteria:

* Patients with previous cardiac surgery, diabetes mellitus, hearing impairment and psychiatric or neurological illness were excluded from this study.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 309 (Actual)
Dates: Start 2016-06-15 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Intraoperative awareness | within the first 24 hours during surgery
  by using a semi-structured in-depth questionnaire (a qualitative method adapted to assess memory development and language level in children to encourage their recall quality and reduce their suggestibility)

SECONDARY OUTCOMES:
Duration of mechanical ventilation | within the first 30 days after surgery
  duration of postoperative mechanical ventilation reported in hours
postoperative cardiac ICU stay | within the first 30 days after surgery
  length of stay in the postoperative cardiac ICU (days)
hospital stay | within the first 30 days after surgery
  length of stay in the hospital (days)
changes from baseline serum cortisol at postoperative period | Within the first 7 days postoperative
  changes from baseline serum cortisol at postoperative period
changes from baseline blood sugar at postoperative period | Within the first 7 days postoperative
  changes from baseline blood sugar at postoperative period
child post-traumatic stress disorder (PTSD) | Within the first 7 days postoperative
  child post-traumatic stress disorder (PTSD) by special scale questionnaire
changes in behavior | Within the first 7 days postoperative
  changes in physiological and psychosocial behaviors of children by questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: sayed abd elshafy, MD, Principal Investigator — associate professor
Locations (1):
- Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided